CLINICAL TRIAL: NCT01157624
Title: Application of Nasal Cannula With Oxygen Versus Air During Eye Surgery Under Local Anaesthetic
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Malaya (Other)
Responsible Party: Tan Siaw Boon, Department of Anaesthesiology, University Malaya
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Health Services Research
Other Study IDs: nasalo2
Record Dates: First submitted 2010-07-05; First posted 2010-07-07 (Estimated); Last update posted 2011-08-17 (Estimated); Status verified 2011-08

CONDITIONS: Hypoxia; Hypercapnia
Keywords: hypoxia or hypercarbia during surgery under the drape
MeSH Terms: conditions — Hypoxia; Hypercapnia | interventions — Oxygen; Resuscitation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- oxygen (Active Comparator)
  Interventions: Drug: oxygen
- air supplement (Placebo Comparator)
  Interventions: Drug: oxygen

INTERVENTIONS:
Drug: oxygen — Subjects who are found to desaturate during treatment with air will be supplement with oxygen
  Other Names: resuscitation for hypoxia
  Arms: oxygen
Drug: oxygen — Subjects who are found to desaturate during treatment with air will be supplement with oxygen
  Other Names: resuscitation for hypoxia
  Arms: air supplement

SUMMARY:
The investigators hypothesize that this new nasal cannula will prevent lack of oxygen as well as reduce rebreathing of carbon dioxide under ophthalmic drapes during eye surgery.

DETAILED DESCRIPTION:
Surgery involvement the eye has widely been done under local anaesthesia provided by the ophthalmologists. Patients are often awake or mildly sedated during the surgery. However, due to the surgical drape which covers the patients face and beyond in order to maintain sterility of the surgical field, it may lead to hypoxia in these patients and retention of exhaled air within the confined space under the drape. This may lead to patient discomfort and the surgeon will face difficulty when the patient becomes restless and unable to be still for the surgery.

Various studies had been conducted using nasal cannula with oxygen or air which is administered to patients having cataract surgery under local anaesthetics and the results has so far been inconclusive.

One study evaluated the saturation of O2 in arterial blood, the partial pressure of O2 in arterial blood (PaO2), the partial pressure of CO2 in arterial blood (PaCO2) and the pH. The operative blood gas parameters were maintained in the air inhalation patients. Oxygen supplement caused significant increase in the saturation of O2 in arterial blood and in PaO2. There was no difference between the two groups in PaCO2. The pH of the arterial blood showed a statistically significant decrease in the patients with O2 supplement. This shift to more acidotic levels could cause central nervous system depression with reduced respiratory stimulus. Recommendation was to administer air rather than O2 to patients during cataract surgery.[1]

Another clinical trials have shown that O2 application by nasal cannula prevents hypoxia but not rebreathing of CO2 in patients undergoing eye surgery under local anaesthetics.[4]

In this clinical trial, we use Duo flow O2 + CO2 sampling cannula designed in a way to deliver O2 and sampling of expired CO2 gases from both nostril simultaneously. The aim of this study is to randomly administer O2 or air through a new nasal cannula to patients undergoing eye surgery under local anaesthetic and to evaluate the significance of O2 supplement and whether CO2 retention has an indirect effect to it.

ELIGIBILITY:
Inclusion Criteria:

* (ASA) physical status I, II or III, adult age 40-80 years old group, scheduled to undergo elective eye surgery under local anaesthetic at UMMC will be enrolled in this study.

Exclusion Criteria:

* pre-existing pulmonary diseases, Psychological disorders, Neurological disorders and patients required sedation.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2010-05; Primary Completion 2010-10 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Evidence of desaturation during intraoperative period under the drape | Intraoperative period

CONTACTS AND LOCATIONS:
Locations (1):
- University Malaya Medical Center, Kuala Lumpur, Federal Teritory, Malaysia